CLINICAL TRIAL: NCT00512525
Title: Intravenous Ghrelin Infusion Decreases Insulin Sensitivity in Healthy Young Men
Brief Title: Ghrelin Decreases Insulin Sensitivity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Esben T. Vestergaard, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: ETV2007
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Ghrelin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Placebo Comparator)
  Interventions: Drug: Ghrelin and saline (as placebo)

INTERVENTIONS:
Drug: Ghrelin and saline (as placebo) — Intravenous infusion

SUMMARY:
Ghrelin administration increases appetite and, in rodents, induces weight gain. The aim of this study is to investigate the effect of short term ghrelin administration to humans on metabolism.

DETAILED DESCRIPTION:
The current study is initiated in order to assess the impact of acute ghrelin administration on insulin resistance measured by a hyperinsulinemic euglycemic clamp. Second, as free fatty acid is the predominant substrate during fasting, we aim to asses the effects of ghrelin on local and systemic lipolysis.

ELIGIBILITY:
Inclusion Criteria:

* healthy men, age >= 18 yr age < 50 yr, body mass index < 27.5 kg/m2above or equal to 18 yr

Exclusion Criteria:

* any disease, use of prescribed medication, age < 18 yr or >= 50 yr

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2003-01; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | End of clamp period

SECONDARY OUTCOMES:
Effects on lipolysis | End of basal and end og clamp period

CONTACTS AND LOCATIONS:
Overall Officials: Ole Schmitz, MD, Study Director — Department of Pharmacology, University of Aarhus, Denmark